CLINICAL TRIAL: NCT04790643
Title: Elaboration and Analysis of a New Cardiac Risk Stratification Protocol Based on Clinical and Physical Variables to Predict the Occurrence of Signs and Symptoms During a Cardiac Rehabilitation Program
Brief Title: Elaboration and Analysis of a New Cardiac Risk Stratification Protocol Based on Clinical and Physical Variables
Status: Completed | Type: Observational
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luiz Carlos Marques Vanderlei, PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Other Study IDs: 35831220.8.0000.5402
Record Dates: First submitted 2021-02-17; First posted 2021-03-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor
Keywords: Cardiac Rehabilitation; Cardiac Risk Stratification; Exercise; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stage 1 - Development of the new cardiac risk stratification protocol: This will be a prospective cohort study, in which individuals attending cardiac rehabilitation programs will be assessed by clinical and physical variables that will be used to guide the elaboration of the cardiac risk stratification protocol. After this initial evaluation, the volunteers will be followed for 2 months during their habitual cardiac rehabilitation routine for the evaluation and registry of the occurrence of minor adverse events, defined as signs and symptoms (arrhythmias, blood pressure alterations, tachypnea, pallor, chest pain, cramps, muscle pain, fatigue, and nausea). The cardiac rehabilitation program in which the volunteers will be recruited is based on moderate-intensity aerobic exercise.
  Interventions: Other: Exercise-based cardiac rehabilitation program (Stage 1)
- Stage 2 - Reproducibility and efficiency of the new protocol: This will be a prospective cohort study, in which a new sample of individuals attending cardiac rehabilitation programs will be assessed by clinical and physical variables and stratified in one of the three following risk classes: "low risk", "moderate risk", and "high risk" accordingly to the new risk stratification protocol. After that, the sample will be followed for 2 months of rehabilitation to the evaluation of the occurrence of signs and symptoms. The cardiac rehabilitation program from where the volunteers will be recruited is based on moderate-intensity aerobic exercise and resistance training. With these data, the reproducibility and efficiency of the protocol will be evaluated.
  Interventions: Other: Exercise-based cardiac rehabilitation program (Stage 2)
- Stage 3 - Protocols´ agreement between evaluators: This will be a cross-sectional observational study in which a new sample of participants will be evaluated by two independent physiotherapists for clinical and physical variables, and based on these data will be stratified by the new protocol by the same evaluators independently. After these procedures, the protocol´s agreement between evaluators will be analyzed.

INTERVENTIONS:
Other: Exercise-based cardiac rehabilitation program (Stage 1) — In Stage 1 the volunteers will perform 24 sessions of exercise-based cardiac rehabilitation. The rehabilitation session is composed of the following activities: I. Initial rest (where the vital signs are evaluated); II. Warming-up (composed of 15 minutes of stretching and global exercises); III. Aerobic exercise (composed of 30 minutes of treadmill or cycle ergometer exercise, the intensity established varies from 40 to 70% of the heart rate reserve for those diagnosed with cardiovascular diseases and from 60 to 80% of the heart rate reserve for those with only cardiac risk factors); IV. Cooldown (composed of 5 minutes of slow walking).
  Groups: Stage 1 - Development of the new cardiac risk stratification protocol
Other: Exercise-based cardiac rehabilitation program (Stage 2) — In Stage 2, the volunteers will perform 24 sessions of exercise-based cardiac rehabilitation. The rehabilitation session is composed of the following activities: I. Initial rest; II. Warming-up; III. Aerobic exercise (these three activities are the same as stage 1); IV. Resistance training (composed of 15 minutes of individualized resistance exercises); V. Cooldown.
  Groups: Stage 2 - Reproducibility and efficiency of the new protocol

SUMMARY:
This research project has as objective the elaboration and analysis of a new cardiac risk stratification protocol based on clinical and physical variables to predict the occurrence of signs and symptoms during a cardiac rehabilitation program. To this aim, the study will be developed in three stages. The first stage consists of a prospective longitudinal observational study, in which participants of exercise-based cardiac rehabilitation will undergo a physiotherapy evaluation in terms of physical and clinical aspects. After this initial assessment, participants will be followed for 2 months of rehabilitation, when the occurrence of signs and symptoms (chest pain, fatigue, dizziness, arrhythmias, and other minor events) during exercise will be recorded. Based on the data from the initial assessment and the occurrence of signs and symptoms a new cardiac risk stratification protocol will be developed. The second stage of this project consists of another prospective longitudinal observational study in which a new sample of individuals attending cardiac rehabilitation programs will be assessed and stratified for the risk of the occurrence of signs and symptoms during exercise by the new protocol developed. After the risk stratification, this sample will be followed for 2 months and the occurrence of signs and symptoms will be recorded. With this data, the reproducibility and efficacy of the protocol will be evaluated. The third stage of this project consists of a cross-sectional observational study, in which a new sample of participants will be evaluated by two independent physiotherapists for clinical and physical variables, and based on these data will be stratified by the new protocol by the same evaluators independently. After these procedures, the protocol´s agreement between evaluators will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Main medical diagnostic of any cardiovascular disease and/or presence of cardiovascular risk factors
* Be participating in exercise-based cardiac rehabilitation

Exclusion Criteria:

* Orthopedic and/or neurologic conditions that preclude the realization of any of the physical and clinical evaluations
* Do not complete 24 cardiac rehabilitation sessions during the follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be recruited from cardiac rehabilitation centers located in Presidente Prudente - SP, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms | Baseline assessment
  The occurrence rate of signs and symptoms will be evaluated during the exercise performed in cardiac rehabilitation programs. The signs and symptoms considered are: arrhythmia, the elevation of systolic and diastolic blood pressure, tachypnea, pallor, angina, cramp, muscle pain, fatigue, and nausea.
Resting heart rate | Baseline assessment
  Evaluated through a heart rate monitor during a resting period of 20 minutes. The mean heart rate obtained between the 5th and 20th minutes will be considered.
Blood pressure | Baseline assessment
  Evaluated indirectly by an experienced physiotherapist using a stethoscope and a sphygmomanometer. The blood pressure will be evaluated three times after a resting period of 15 minutes. The mean value of the last 2 measures will be considered.
Maximum inspiratory pressure | Baseline assessment
  Evaluated through a manovacuometer. This assessment will be evaluated three times and the value considered will be the mean of all measures.
Maximum expiratory pressure | Baseline assessment
  Evaluated through a manovacuometer. This assessment will be evaluated three times and the value considered will be the mean of all measures.
Peak expiratory flow | Baseline assessment
  Evaluated through the spirometric examination performed by an experienced physiotherapist.
Forced expiratory volume in the first second | Baseline assessment
  Evaluated through the spirometric examination performed by an experienced physiotherapist.
Forced vital capacity | Baseline assessment
  Evaluated through the spirometric examination performed by an experienced physiotherapist.
Cardiac autonomic modulation - RMSSD index | Baseline assessment
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. To obtain the RR intervals time series, the volunteer will rest for 30 minutes in spontaneous breathing. Will be considered 1000 consecutive RR intervals recorded between the 5th and 30th minutes of rest. The RMSSD index corresponds to the root-mean square of differences between adjacent normal RR intervals in a time interval, expressed in milliseconds.
Cardiac autonomic modulation - SDNN index | Baseline assessment
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. To obtain the RR intervals time series, the volunteer will rest for 30 minutes in spontaneous breathing. Will be considered 1000 consecutive RR intervals recorded between the 5th and 30th minutes of rest. The SDNN index corresponds to the standard deviation of all normal RR intervals recorded in a time interval, expressed in milliseconds.
Cardiac autonomic modulation - LF index (ms²) | Baseline assessment
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. To obtain the RR intervals time series, the volunteer will rest for 30 minutes in spontaneous breathing. Will be considered 1000 consecutive RR intervals recorded between the 5th and 30th minutes of rest. The LF index is the low-frequency component of the oscillatory components of heart rate variability, and ranges from 0.04 to 0.15 Hz.
Cardiac autonomic modulation - HF index (ms²) | Baseline assessment
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. To obtain the RR intervals time series, the volunteer will rest for 30 minutes in spontaneous breathing. Will be considered 1000 consecutive RR intervals recorded between the 5th and 30th minutes of rest. The HF index is the high-frequency component of the oscillatory components of heart rate variability, and ranges from 0.15 to 0.4 Hz.
Cardiac autonomic modulation - LF index (nu) | Baseline assessment
  The LF index expressed in normalizefd units (nu) is obtained by dividing the power in milliseconds by the total power spectrum, minus the very low frequency component and multiplied by 100.
Cardiac autonomic modulation - HF index (nu) | Baseline assessment
  The HF index expressed in normalizefd units (nu) is obtained by dividing the power in milliseconds by the total power spectrum, minus the very low frequency component and multiplied by 100.
Cardiac autonomic modulation - LF/HF ratio | Baseline assessment
  This index is obtained by dividing the LF (ms²) value by the HF (ms²) value.
Cardiac autonomic modulation - SD1 index | Baseline assessment
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. To obtain the RR intervals time series, the volunteer will rest for 30 minutes in spontaneous breathing. Will be considered 1000 consecutive RR intervals recorded between the 5th and 30th minutes of rest. The SD1 index corresponds to the dispersion of points perpendicular to the line of identity of the ellipse obtained from the Poincaré plot. Expressed in milliseconds.
Cardiac autonomic modulation - SD2 index | Baseline assessment
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. To obtain the RR intervals time series, the volunteer will rest for 30 minutes in spontaneous breathing. Will be considered 1000 consecutive RR intervals recorded between the 5th and 30th minutes of rest. The SD1 index corresponds to the dispersion of points along the line of identity of the ellipse obtained from the Poincaré plot. Expressed in milliseconds.
Cardiac autonomic modulation - SD1/SD2 ratio | Baseline assessment
  This index is obtained by dividing the SD1 value by the SD2 value.
Quadriceps muscle strength | Baseline assessment
  Evaluated through a digital dynamometer. The volunteer will perform three maximal isometric contractions of quadriceps with a duration of 5 seconds. The value considered will be the higher one among the three contractions.
Submaximal functional capacity | Baseline assessment
  Evaluated by the 6-minute walk test. The values considered will be the distance covered and the % of the predicted value reached.
Body mass index | Baseline assessment
  Calculated using the data of body mass assessed by a digital scale and height evaluated through a stadiometer.
Waist circumference | Baseline assessment
  Measured with an inelastic measuring tape at the lower abdominal perimeter. Three measurements will be taken and the average of the values obtained will be considered.
Abdominal circumference | Baseline assessment
  Measured with an inelastic measuring tape at the umbilical scar line. Three measurements will be taken and the average of the values obtained will be considered.
Hip circumference | Baseline assessment
  Measured with an inelastic measuring tape at the largest perimeter in the gluteal region. Three measurements will be taken and the average of the values obtained will be considered.
Arm circumference | Baseline assessment
  Measured with an inelastic measuring tape at the midpoint between the acromion and the olecranon with the upper limb relaxed. Three measurements will be taken and the average of the values obtained will be considered.
Calf circumference | Baseline assessment
  Measured with an inelastic measuring tape at the largest circumference in the region of the right calf with the lower limb relaxed without receiving weight. Three measurements will be taken and the average of the values obtained will be considered.
Basal metabolic rate (cal/day) | Baseline assessment
  Evaluated through a tetrapolar electrical bioimpedance examination.
Total body water (%) | Baseline assessment
  Evaluated through a tetrapolar electrical bioimpedance examination.
Total water in the lean mass (%) | Baseline assessment
  Evaluated through a tetrapolar electrical bioimpedance examination.
Resistance (Ohms) | Baseline assessment
  Evaluated through a tetrapolar electrical bioimpedance examination.
Reactance (Ohms) | Baseline assessment
  Evaluated through a tetrapolar electrical bioimpedance examination.
Body fat (%) | Baseline assessment
  Evaluated through a tetrapolar electrical bioimpedance examination.
Body fat (Kg) | Baseline assessment
  Evaluated through a tetrapolar electrical bioimpedance examination.
Total lean mass (Kg) | Baseline assessment
  Evaluated through a tetrapolar electrical bioimpedance examination.

OTHER OUTCOMES:
Reproducibility of the risk stratification protocol to predict the signs and symptoms occurrence | Through study completion, an average of 2 years
  The agreement between the risk class and the number of signs and symptoms that occurred will be calculated using the Kappa intraclass correlation coefficient.
Efficacy of the risk stratification protocol to predict the signs and symptoms occurrence | Through study completion, an average of 2 years
  The effectiveness of the protocol in predicting the occurrence of signs and symptoms will be assessed by analyzing the ROC curve, by measuring sensitivity, specificity and area under the curve (AUC).
Agreement between evaluators | Through study completion, an average of 2 years
  Reliability between evaluators will be assessed using the percentage of agreement and disagreement and the Kappa index.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos Marques Vanderlei, PhD, Principal Investigator — Universidade Estadual Paulista "Julho de Mesquita Filho" (UNESP)
Locations (1):
- Universidade Estadual Paulista Júlio de Mesquita Filho, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided